CLINICAL TRIAL: NCT00689143
Title: A Phase I, Open-Label, Single Center, Safety/Tolerability and Pharmacokinetic Study of Leukine® Administrated in the Gingiva as Three Single Doses on Separate Days
Brief Title: A Safety/Tolerability and Pharmakokinetic Study of Sargramostim Administrated in the Gingiva
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innoventus Project AB (Industry)
Collaborators: Uppsala University (Other)
Responsible Party: Innoventus Project AB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPPIS-0604
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sargramostim
  Other Names: GM-CSF; Leukine

SUMMARY:
This exploratory study is the first study in a clinical program where the overall objective is to develop a novel pharmaceutical therapy comprising local administration of GM-CSF for the treatment of periodontitis. The project hypothesis is based on GM-CSF's antibacterial and putative bone regeneration properties. Periodontitis is the major cause of tooth loss in people over 35 years of age. An effective pharmacological treatment is today lacking and the actual therapy would represent a new treatment option for the large patient group suffering from the disease.

DETAILED DESCRIPTION:
It is suggested that local administration of GM-CSF in the gingival tissue next to the periodontal destruction may reduce the infectious condition by an antibacterial effect via stimulation of neutrophil phagocytosis of bacteria, enhanced functional activities of monocytes and granulocytes, as well as stimulation of bone tissue recalcification.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals (male or female) referred to Dept of Oral & Maxillofacial surgery to have a lower wisdom tooth surgically extracted
* ≥ 20 and ≤ 40 years of age
* Analysis results of blood status within normal reference ranges
* Ability to attend the scheduled visits for evaluation procedures
* Women with child-bearing potential: use of an adequate method of contraception to avoid pregnancy throughout the study
* Signed informed consent

Exclusion Criteria:

* Any significant disease (acute or chronic) or any medication with concomitant oral manifestations that in the opinion of the investigator would interfere with safety evaluation of Leukine.
* An active osseous infection or periodontal infection, any active mucosal lesions or a history of acute necrotizing ulcerative gingivitis.
* Current use of anti-coagulant therapy or within 10 days from baseline
* Current use of immunomodulating medication
* Current use of corticosteroids (Amendment 1: topical use permitted).
* Current use of lithium.
* Use of tobacco products or nicotine replacement therapy
* Alcohol or drug abuse
* HIV or hepatitis infection
* Pregnancy or lactation
* Participation in another clinical study on medicinal products at the time of inclusion
* Lack of suitability for participation in the trial, for any reason, as judged by the Investigator.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To establish the safety profile of three escalating doses of Leukine when given as single intragingival injections on separate days

SECONDARY OUTCOMES:
To perform a pharmacokinetic evaluation after administration of three escalating doses of Leukine into the gingival tissue as single doses on separate days

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hirsch, Prof., Principal Investigator — Dept of Oral & Maxillofacial Surgery, Uppsala University Hospital, Sweden
Locations (1):
- Dept of Oral & Maxillofacial Surgery, Uppsala, Sweden